CLINICAL TRIAL: NCT02632448
Title: A Phase 1b/2a Three-Part Open-Label Multicenter Study to Evaluate the Safety and Efficacy of LY2880070 as Monotherapy and in Combination With Gemcitabine in Patients With Advanced or Metastatic Cancer
Brief Title: A Study of LY2880070 in Participants With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Esperas Pharma Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ESPS-001
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors; Colorectal Cancer; Breast Cancer; Ovarian Cancer; Colon Cancer; Rectal Cancer; Neoplasms; Endometrial Cancer; Soft Tissue Sarcoma; Triple Negative Breast Cancer; Pancreas Cancer; Pancreatic Cancer
Keywords: Metastatic cancer; Advanced cancer; Recurrent cancer; Colorectal neoplasms; Triple negative breast cancer; Ovarian neoplasms; Colon neoplasms; Rectal neoplasms; Triple negative breast neoplasms; Gastrointestinal stromal tumor; Pancreatic Neoplasms; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasms; Endometrial Neoplasms; Sarcoma; Triple Negative Breast Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Recurrence; Gastrointestinal Stromal Tumors | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A: LY2880070 (Experimental): Multiple oral doses of LY2880070 during 21-day cycles
  Interventions: Drug: LY2880070
- Part A: LY2880070 with Gemcitabine (Experimental): Multiple oral doses of LY2880070, and Gemcitabine administered intravenously during 21-day cycles
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part A: LY2880070 (Metabolism Phenotype) (Experimental): Multiple oral doses of LY2880070 administered during 21 day cycles, to participants who are poor metabolizers
  Interventions: Drug: LY2880070
- Part B: LY2880070 and Gemcitabine (Breast) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part B: LY2880070 and Gemcitabine (Colorectal) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part B:LY2880070 and Gemcitabine (Ovarian) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part B: LY2880070 and Gemcitabine (Endometrial) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part B: LY2880070 and Gemcitabine (Soft Tissue Sarcoma (STS)) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part B: LY2880070 and Gemcitabine (Pancreatic) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine
- Part C: LY2880070 and Gemcitabine (High Grade Serous Ovarian Cancer) (Experimental): Multiple oral doses of LY2880070 during 21-day cycles with Gemcitabine (administered intravenously)
  Interventions: Drug: LY2880070; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2880070 — Capsules
Drug: Gemcitabine — 50 to 600 milligrams per square meter of body surface area (mg/m2)
  Other Names: Gemzar
  Arms: Part A: LY2880070 with Gemcitabine; Part B: LY2880070 and Gemcitabine (Breast); Part B: LY2880070 and Gemcitabine (Colorectal); Part B: LY2880070 and Gemcitabine (Endometrial); Part B: LY2880070 and Gemcitabine (Pancreatic); Part B: LY2880070 and Gemcitabine (Soft Tissue Sarcoma (STS)); Part B:LY2880070 and Gemcitabine (Ovarian); Part C: LY2880070 and Gemcitabine (High Grade Serous Ovarian Cancer)

SUMMARY:
The main purpose of this 3-part study is to evaluate the safety and efficacy of the study drug known as LY2880070 in participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have an estimated life expectancy of greater than or equal to (≥)12 weeks
* Have adequate organ function
* Have received 1-4 prior systemic therapies for locally advanced or metastatic disease
* Agree to use medically approved contraceptives during the study and for 3 months following the last study treatment
* All females must have a negative serum pregnancy test result, and females of child-bearing potential must have a negative urine pregnancy test result, prior to the first study treatment
* Have tumor lesions considered measurable by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Must be, in the judgment of the investigator, an appropriate candidate for experimental therapy, and no standard therapy would confer clinical benefit

For Part A

* Must have evidence of cancer (solid tumors, excluding glioblastoma and primary brain tumor) that is advanced or metastatic
* For the Metabolism Phenotype Arm in Part A, participants must have a Cytochrome P450 (CYP2D6) poor metabolizer phenotype

For Part B

* Have advanced or metastatic colorectal cancer, triple negative breast cancer (per American Society of Clinical Oncology-College of American Pathology guidelines), epithelial ovarian cancer, endometrial, soft tissue sarcoma, pancreatic cancer

  * For TNBC:

    * Recurrent/refractory Triple Negative Breast Cancer (TNBC) defined as any beast cancer that expresses <1% estrogen receptor (ER) and <1% progesterone receptor (PR) and is Her2 negative
  * For Colorectal (CRC):

    * Must have histologically confirmed advanced or metastatic colorectal cancer
  * For Ovarian Cancer:

    * Must have histologically confirmed advanced or metastatic epithelial ovarian cancer
    * Must be eligible to receive Gemzar (GEM) and not refractory to GEM/carboplatin
    * Must have the ability to tolerate GEM
    * May have received GEM as previous therapy
  * For Endometrial cancer:

    * Must have histologically confirmed endometrial cancer that is metastatic or locally advanced
    * Must have failed at least 1 prior chemotherapy
  * For STS:

    * Must have histologically confirmed STS that is metastatic or locally advanced
    * Patients with gastrointestinal stromal tumors (GIST) must have failed a KIT inhibitor
    * Must have failed at least 1 prior chemotherapy
  * For Pancreatic Cancer:

    * Must have histologically confirmed pancreatic cancer that is metastatic or locally advanced
    * Must have failed at least 1 prior chemotherapy regimen
  * For Part C
  * Participants with high grade serous ovarian cancer (HGSOC) will be screened for specific genetic signatures

Exclusion Criteria:

* Have received treatment with an investigational drug which has not received regulatory approval within 21 days of first study treatment
* Have symptomatic central nervous system (CNS) metastasis
* Females who are pregnant or nursing
* Have known positive test results of human immunodeficiency virus, or have chronic active hepatitis A, B or C
* Have a corrected QT interval (QTcB) greater than (>) 470 milliseconds (msec) (female) or >450 msec (male), or a history of congenital long QT syndrome
* Have had a bone marrow transplant
* Have participated in this study, or are currently enrolled in another clinical study of an investigational medicinal product
* Have had radiation therapy to >25% of bone marrow
* For Part B

  * Have a history of another active cancer within the past year, except cervical cancer in situ, in situ carcinoma of the bladder, basal cell carcinoma of the skin, or another in situ carcinoma that is considered cured

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Estimated)
Dates: Start 2016-05-16 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(s) | Baseline through Cycle 1 (Estimated up to 21 days)

SECONDARY OUTCOMES:
Number of dose limiting toxicities (DLTs) | Baseline through Cycle 1 (Estimated up to 21 days)
Area under the plasma concentration versus time curve from time zero to 24 hours post-dose (AUC0-24) | Baseline to 24-hours post dose (up to Day 20 in Cycle 1)
Peak plasma concentration (Cmax) | Baseline to 24 hours post-dose (up to Day 20 in Cycle 1)
Time to reach maximum plasma concentration (tmax) | Baseline to 24 hours post dose (up to Day 20 in Cycle 1)
Change from baseline in white blood cell count | Baseline to 24 hours post dose (up to Day 20 in Cycle 1)
Change from baseline in neutrophil count | Baseline to 24 hours post dose (up to Day 20 in Cycle 1)
Change from baseline in lymphocyte count | Baseline to 24 hours post dose (up to Day 20 in Cycle 1)
Number of participants with tumor response (objective response rate) as measured by the Response Evaluable Criteria in Solid Tumors (RECIST v.1.1) | Baseline to study completion (estimated up to 4 years)
Duration of objective response | Baseline to study completion (estimated up to 4 years)
Best response | Baseline to study completion (estimated up to 4 years)
Progression free survival | Baseline to study completion (estimated up to 4 years)
Overall survival | Baseline up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Email: Darcy.Vincett@ozmosisresearch.ca, Study Director — Esperas Pharma Inc.
Locations (16):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - University Health Network - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Croatia (2):
  - General Hospital Zadar, Zadar
  - University Hospital Centre Zagreb, Zagreb
- Poland (4):
  - Centrum Onkologii im. prof. F. Łukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne Osrodek Badan Klinicznych Wczesnych Faz, Gdansk
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o. o., Krakow
  - Szpital Specjalistyczny im. L. Rydygiera w Krakowie sp. z o. o., Krakow

REFERENCES:
- [Result] W.H. Miller, A.F. Shields, D. Provencher, L. Gilbert, G. Shapiro, A.M. Oza, J. Spratlin, S. Lheureux, G. Bhat, S. Salvador, P. Nunes, S. Lau, I. Weiner, J. Keene, S. Zaknoen, P. Smith, J. Stille, D. Vincett, Q.S-C. Chu, 537P A phase I/II study of oral chk1 inhibitor LY2880070 in combination with low-dose gemcitabine in patients with advanced or metastatic ovarian cancer, Annals of Oncology, Volume 33, Supplement 7, 2022, Pages S793-S794, ISSN 0923-7534, https://doi.org/10.1016/j.annonc.2022.07.665. (https://www.sciencedirect.com/science/article/pii/S0923753422025169)
- [Result] DOI: 10.1200/JCO.2020.38.15_suppl.3579 Journal of Clinical Oncology 38, no. 15_suppl (May 20, 2020) 3579-3579.
- [Result] DOI: 10.1200/JCO.2020.38.15_suppl.3581 Journal of Clinical Oncology 38, no. 15_suppl (May 20, 2020) 3581-3581.
- [Derived] Huffman BM, Feng H, Parmar K, Wang J, Kapner KS, Kochupurakkal B, Martignetti DB, Sadatrezaei G, Abrams TA, Biller LH, Giannakis M, Ng K, Patel AK, Perez KJ, Singh H, Rubinson DA, Schlechter BL, Andrews E, Hannigan AM, Dunwell S, Getchell Z, Raghavan S, Wolpin BM, Fortier C, D'Andrea AD, Aguirre AJ, Shapiro GI, Cleary JM. A Phase I Expansion Cohort Study Evaluating the Safety and Efficacy of the CHK1 Inhibitor LY2880070 with Low-dose Gemcitabine in Patients with Metastatic Pancreatic Adenocarcinoma. Clin Cancer Res. 2023 Dec 15;29(24):5047-5056. doi: 10.1158/1078-0432.CCR-23-2005. PMID 37819936